CLINICAL TRIAL: NCT06560190
Title: Orthopaedic Manual Physical Therapy as Part of the Postpartum Care Continuum for Active-Duty Service Members
Brief Title: Orthopaedic Manual Physical Therapy as Part of the Postpartum Care Continuum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Casey Shutt-Hoblet, MAJ Casey Shutt-Hoblet, PT, DPT, Brooke Army Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT4Postpartum
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Postpartum; Pregnancy Related
Keywords: Postpartum; Physical Activity; Pregnancy; Service Member; Physical Therapy
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postpartum Study Participant (Experimental): Pragmatic Orthopaedic Physical Therapy
  Interventions: Other: Orthopaedic Manual Physical Therapy

INTERVENTIONS:
Other: Orthopaedic Manual Physical Therapy — Individualized Treatment

SUMMARY:
Data shows us that injury risk increases in the first year postpartum. There is a paucity of literature regarding MSK injuries in postpartum military women. A unique challenge that postpartum service members face is the increased stress of training for and having to pass a physical fitness test directly tied to their career advancement.

While there is epidemiological data across multiple branches of service, there is a gap in the literature in terms of how to appropriately address these decreased fitness levels and better understand the root causes. American College of Gynecology (ACOG) recommends that the postpartum visit include actionable information on return to physical activity. However, a large majority of women report receiving no guidance on how to engage in physical activity during pregnancy and in the postpartum period.

Physical therapy is commonly used to help individuals return to physical activity following orthopaedic surgeries, but it is not frequently utilized to assist the postpartum population in progressing back to physical activity. Orthopaedic Manual Physical Therapists (OMPTs) are uniquely trained to address musculoskeletal symptoms and progress physical activity. An OMPT evaluation and treatment could facilitate increased physical activity and improve health-related quality of life, supporting the ACOG recommendation to make postpartum care an ongoing multidisciplinary process.

DETAILED DESCRIPTION:
The purpose of this study is to 1) Describe changes in health-related quality of life in postpartum women following eight weeks of orthopaedic physical therapy management as part of the postpartum care continuum for active-duty service members 2) Describe changes in pain and physical activity levels following eight-weeks of OMPT management in this same sample and 3) Determine whether select patient characteristics associated with improvement physical function scores following this same eight-week program of OMPT.

This is a Quasi-experimental one-group repeated measures study. Participants who meet the inclusion criteria will be evaluated by board certified orthopedic physical therapist who is a fellow-in-training.The initial evaluation and treatment will be provided over an 8 week period with a minimum of 3 visits. The treatment approach will be initiated at the initial visit and will be based on standard of care OMPT treatment and existing rehab frameworks for postpartum pelvic girdle pain, low back pain and return to physical activity.

At the 8-week time point, participants will complete final outcomes tools. Participants will be discharged from the study, but they can choose to continue physical therapy intervention with their treating provider if they desire. Data beyond the 8-week mark will not be saved for the research trial.

ELIGIBILITY:
Inclusion Criteria:

* Female Active-Duty Service Member
* Postpartum >6 weeks and <6 months
* Cleared by OBGYN at postpartum follow-up to initiate physical activity

Exclusion Criteria:

* Current or ongoing treatment by an orthopaedic physical therapist
* Separating from military service in the next 6 months
* Current permanent profile for a musculoskeletal condition
* Peripartum Hysterectomy

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-07-05 (Estimated); Study Completion 2025-07-05 (Estimated)

PRIMARY OUTCOMES:
36-Item Short Form Survey Instrument (SF36) | Baseline, 4 weeks and 8 weeks
  The 36-Item Short Form Survey Instrument (SF 36) is the most widely used quality of life tool in the postpartum population. The lowest score on each subscale is zero and the highest score on each subscale is 100. A higher score is better.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire- Short Form (IPAQ) | Baseline, 4 weeks and 8 weeks
  We will use the International physical activity questionnaire short form to assess physical activity level. The lowest score is zero and the highest score is not identified although scores over 16 hours of physical activity per day should be excluded as an outlier. A higher score is better.
Numeric Pain Rating Scale (NPRS) | Baseline, 4 weeks and 8 weeks
  The Numeric Pain Rating Scale (NPRS) will be used to measure pain.The lowest score is 0 and the highest score is 10. A lower score is better.
Cozean Pelvic Dysfunction Screening Protocol | Baseline, 4 weeks and 8 weeks
  Orthopaedic physical therapists should utilize the Cozean protocol to screen which patients need a pelvic floor rehab referral following the DHA practice recommendation for Pelvic Health and Postpartum Rehabilitation Services. The lowest score is zero and highest score is 10. A higher score does not indicate more dysfunction. A cutoff of 3 is applied to indicate a referral is needed for pelvic floor physical therapy.
Edinburgh Postnatal Depression Scale (EPDS) | Baseline
  This tool will be used in accordance with the DHA Practice Recommendation for Behavioral Health Screening and Referral in Pregnancy and Postpartum at the initial evaluation to screen for depression in postpartum patients. The lowest score is zero and highest score is thirty. A higher score is worse and indicates need for behavioral health referral.

CONTACTS AND LOCATIONS:
Overall Officials: Casey Shutt-Hoblet, DPT, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Will consider dissemination on a case by case basis.

REFERENCES:
- [Background] Iobst SE, Smith DC, Best NI, Allard RJ, Trego LL. A Scoping Review of Pregnancy, Childbirth, and the Postpartum Period in Active Duty U.S. Military Women. Womens Health Issues. 2021 Aug 25;31 Suppl 1:S81-S92. doi: 10.1016/j.whi.2020.05.005. PMID 34454706
- [Background] Miller MJ, Kutcher J, Adams KL. Effect of Pregnancy on Performance of a Standardized Physical Fitness Test. Mil Med. 2017 Nov;182(11):e1859-e1863. doi: 10.7205/MILMED-D-17-00093. PMID 29087853
- [Background] Weina SU. Effects of pregnancy on the Army Physical Fitness Test. Mil Med. 2006 Jun;171(6):534-7. doi: 10.7205/milmed.171.6.534. PMID 16808137
- [Background] DeGroot DW, Sitler CA, Lustik MB, Langan KL, Hauret KG, Gotschall MH, Gehrich AP. The effect of pregnancy and the duration of postpartum convalescence on the physical fitness of healthy women: A cohort study of active duty servicewomen receiving 6 weeks versus 12 weeks convalescence. PLoS One. 2021 Jul 28;16(7):e0255248. doi: 10.1371/journal.pone.0255248. eCollection 2021. PMID 34320030
- [Background] Armitage NH, Smart DA. Changes in Air Force fitness measurements pre- and post-childbirth. Mil Med. 2012 Dec;177(12):1519-23. doi: 10.7205/milmed-d-12-00248. PMID 23397699
- [Background] ACOG Committee Opinion No. 736: Optimizing Postpartum Care. Obstet Gynecol. 2018 May;131(5):e140-e150. doi: 10.1097/AOG.0000000000002633. PMID 29683911
- [Background] Doran F, Davis K. Factors that influence physical activity for pregnant and postpartum women and implications for primary care. Aust J Prim Health. 2011;17(1):79-85. doi: 10.1071/PY10036. PMID 21616029
- [Background] Selman R, Early K, Battles B, Seidenburg M, Wendel E, Westerlund S. Maximizing Recovery in the Postpartum Period: A Timeline for Rehabilitation from Pregnancy through Return to Sport. Int J Sports Phys Ther. 2022 Oct 1;17(6):1170-1183. doi: 10.26603/001c.37863. eCollection 2022. PMID 36237644
- [Background] Christopher, S.M., et al., Rehabilitation of the Postpartum Runner: A 4-Phase Approach. Journal of Women's Health Physical Therapy, 2022. 46(2): p. 73-86.